CLINICAL TRIAL: NCT01460940
Title: A Phase II Trial of Panobinostat and Lenalidomide in Patients With Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Celgene (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-10049; NCI-2011-03323 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2011-10-14; First posted 2011-10-27 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Adult Lymphocyte Depletion Hodgkin Lymphoma; Adult Lymphocyte Predominant Hodgkin Lymphoma; Adult Mixed Cellularity Hodgkin Lymphoma; Adult Nodular Lymphocyte Predominant Hodgkin Lymphoma; Adult Nodular Sclerosis Hodgkin Lymphoma; Recurrent Adult Hodgkin Lymphoma
Keywords: refractory Hodgkin's lymphoma; panobinostat; lenalidomide
MeSH Terms: conditions — Hodgkin Disease | interventions — Panobinostat; Histone Deacetylase Inhibitors; Hydroxamic Acids; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide and Panobinostat (Experimental): In the phase I trial, three patients will be enrolled at each dose level, starting at dose level 1 using a standard 3 + 3 dose escalation phase I design.
  Interventions: Drug: panobinostat; Drug: lenalidomide

INTERVENTIONS:
Drug: panobinostat — Administered orally Monday, Wednesday, Friday of every week for 4 weeks. A cycle is define as 28 days.
  Other Names: HDAC inhibitor; LBH589; hydroxamic acid
Drug: lenalidomide — Lenalidomide will be administered orally daily on days 1-21. Lenalidomide will not be given on days 22-28. A cycle is define as 28 days.
  Other Names: CC-5013; Revlimid

SUMMARY:
This phase II trial studies how well giving panobinostat together with lenalidomide works in treating patients with relapsed or refractory Hodgkin lymphoma. Panobinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Giving panobinostat together with lenalidomide may be an effective treatment for Hodgkin lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Determine the overall response rate (ORR), including complete responses (CR) and partial responses (PR), with combined lenalidomide and panobinostat in patients with relapsed or refractory Hodgkin's lymphoma. SECONDARY OBJECTIVES: I. Assess the safety and tolerability of combined lenalidomide and panobinostat in patients with previously treated Hodgkin's lymphoma. II. Determine progression-free survival (PFS) in patients with previously treated Hodgkin's lymphoma receiving combined lenalidomide and panobinostat. III. Evaluate changes in natural killer (NK) cell number and function, plasma cytokines, gene expression profile of peripheral blood, and plasma proteins via proteomics, before, during, and after lenalidomide and panobinostat therapy. IV. Determine levels of histone acetylation before and after treatment with panobinostat. V. Determine the pharmacokinetics of lenalidomide in the presence of panobinostat. VI. To collect deoxyribonucleic acid (DNA) samples for potential later analysis of associations between outcomes and polymorphisms in genes coding for drug metabolizing enzymes, transporters and molecular targets of lenalidomide or panobinostat. OUTLINE: Patients receive panobinostat orally (PO) on days 1, 3, and 5 of weeks 1-4 and lenalidomide PO on days 1-7 of weeks 1-3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up at least every 3 months for 2 years, and then every 6 months for 3-5 years

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed classical or lymphocyte predominant Hodgkin's lymphoma that is relapsed or refractory after at least one prior chemotherapy; patients with Hodgkin's lymphoma may have one of the following World Health Organization (WHO) subtypes:

  * Nodular sclerosis Hodgkin's lymphoma
  * Mixed cellularity Hodgkin's lymphoma
  * Lymphocyte-rich Hodgkin's lymphoma
  * Lymphocyte-deplete Hodgkin's lymphoma
  * Nodular Lymphocyte-predominant Hodgkin's lymphoma
* Patients must have relapsed or progressed after at least one prior cytotoxic chemotherapy

  * Previous autologous or allogeneic stem cell transplantation is permitted
  * Previous treatment with either single agent panobinostat or lenalidomide is permitted
* Absolute neutrophil count (ANC) >= 1200/μL
* Platelets >= 100,000/μl
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit normal (ULN)
* Serum bilirubin =< 1.5 x ULN
* Calculated creatinine clearance >= 60ml/min by Cockcroft-Gault estimation of CrCI
* Measurable Disease must be present either on physical examination or imaging studies; non-measurable disease alone is not acceptable; any tumor mass > 1 cm is acceptable; lesions that are considered non-measurable include the following:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Inflammatory breast disease
  * Lymphangitis cutis/pulmonis
  * Bone marrow involvement (involvement by non-Hodgkin lymphoma should be noted)
* Baseline multi gated acquisition (MUGA) or echocardiogram (ECHO) must demonstrate left ventricular ejection fraction (LVEF) >= 45%
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Able to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to starting Cycle 1 of lenalidomide (prescriptions must be filled within 7 days as required by RevAssist) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant of aspirin or at increased risk of venous thrombosis may use warfarin or low molecular weight heparin)

Exclusion Criteria:

* Patients who are candidates for high dose chemotherapy and autologous stem cell transplantation with curative intent should not be enrolled
* Patients with active central nervous system (CNS) lymphoma
* Use of valproic acid for any medical condition while receiving protocol treatment or within 5 days prior to first panobinostat dose
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

  * History or presence of sustained ventricular tachyarrhythmia; (patients with a history of atrial arrhythmia are eligible but should be discussed with Novartis prior to enrollment)
  * Any history of ventricular fibrillation or Torsade de Pointes
  * Bradycardia defined as heart rate (HR) < 50 beats per minute (bpm); patients with pacemakers are eligible if HR >= 50 bpm
  * Screening electrocardiogram (ECG) with a QTc > 450 msec
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Patients with myocardial infarction or unstable angina =< 6 months prior to starting study drug
  * Other clinically significant heart disease (e.g., congestive heart failure [CHF] New York [NY] Heart Association class III or IV, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat
* Patients with diarrhea > Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Known hypersensitivity to thalidomide or lenalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Pregnant or breastfeeding females
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis B or C; baseline testing for HIV and hepatitis C is not required. Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Concurrent use of other anti-cancer agents or treatments
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10-13; Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Washington University, St Louis, Missouri
  - The Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Maly JJ, Christian BA, Zhu X, Wei L, Sexton JL, Jaglowski SM, Devine SM, Fehniger TA, Wagner-Johnston ND, Phelps MA, Bartlett NL, Blum KA. A Phase I/II Trial of Panobinostat in Combination With Lenalidomide in Patients With Relapsed or Refractory Hodgkin Lymphoma. Clin Lymphoma Myeloma Leuk. 2017 Jun;17(6):347-353. doi: 10.1016/j.clml.2017.05.008. Epub 2017 May 22. PMID 28622959
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide and Panobinostat
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide and Panobinostat
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 45 [22 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Determine the Overall Response Rate (ORR), Including Complete Responses (CR) and Partial Responses (PR)
Description: Overall response rate (CR + PR) will be determined using the International response criteria with combined panobinostat and lenalidomide in patients with relapsed or refractory Hodgkin's lymphoma.
Time Frame: up to 24 months
Measure: Number; unit: percentage of patients
Arm/Group | Lenalidomide and Panobinostat
Number analyzed (Participants) | 24
percentage of patients | 16.7

2. Secondary Outcome: Assess the Safety and Tolerability of Combined Lenalidomide and Panobinostat in Patients With Previously Treated Hodgkin's Lymphoma.
Description: Safety and tolerability will be assessed for patients using the NIH-NCI Common Terminology Criteria (CTCAE) version 4.0
Time Frame: up to 24 months
Population: Grade 3-4 toxicities
Measure: Number; unit: percentage of patients
Arm/Group | Lenalidomide and Panobinostat
Number analyzed (Participants) | 24
percentage of patients
  neutropenia | 58.3
  thrombocytopenia | 41.7
  febrile neutropenia | 25.0
  hypophosphatemia | 25.0

3. Secondary Outcome: Progression-free Survival in Patients With Previously Treated Hodgkin's Lymphoma Receiving Combined Lenalidomide and Panobinostat
Description: Determined from the date of start of therapy to death from any cause or censored at the last date the patient is known to be alive
Time Frame: 3-5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Panobinostat
Number analyzed (Participants) | 24
months | 3.8 [1.8 to 5.9]

ADVERSE EVENTS:
Arm/Group | Lenalidomide and Panobinostat
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 17/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Panobinostat (N=24)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Fatigue (Investigations) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 4 (4)
Infection without Neutropenia (Infections and infestations) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 1 (1)
Hyperbilirubinemia/Transaminitis (Metabolism and nutrition disorders) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Panobinostat (N=24)
Neutropenia (Infections and infestations) | 11 (11)
Lymphopenia (Investigations) | 6 (6)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hyperbilirubinemia/Transaminitis (Metabolism and nutrition disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
Infection without Neutropenia (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No